CLINICAL TRIAL: NCT02241967
Title: Dose Dependent Effects of tDCS on Post-Operative Pain
Acronym: tDCS-TKA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-005-13F; CX001078 (Other Grant/Funding Number: Charleston CSR&D)
Record Dates: First submitted 2014-09-02; First posted 2014-09-16 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Total Knee Arthroplasty (Postoperative Pain); Total Hip Arthroplasty(Postoperative Pain)
Keywords: total knee arthroplasty; pain; post-surgical pain; opioid; transcranial direct current stimulation; tDCS; brain stimulation; total hip arthroplasty; TKA; THA
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- tDCS Full Dose (Experimental): 4 active treatments
  Interventions: Device: 4 Real sessions of Transcranial Direct Current Stimulation
- tDCS Half Dose (Experimental): 2 active treatments
  Interventions: Device: 2 Real Sessions of Transcranial Direct Current Stimulation
- tDCS Minimal dose (Experimental): 1 active treatment
  Interventions: Device: 1 Real Session of Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): no active treatments
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: 4 Real sessions of Transcranial Direct Current Stimulation — Stimulation of brain areas associated with pain perception using low amplitude direct current of 2mA delivered by electrodes attached to the scalp.
  Other Names: tDCS Full Dose
  Arms: tDCS Full Dose
Device: 2 Real Sessions of Transcranial Direct Current Stimulation — Stimulation of brain areas associated with pain perception using low amplitude direct current of 2mA delivered by electrodes attached to the scalp. 2 real sessions of tDCS and 2 sham.
  Other Names: tDCS Half Dose
  Arms: tDCS Half Dose
Device: 1 Real Session of Transcranial Direct Current Stimulation — Stimulation of brain areas associated with pain perception using low amplitude direct current of 2mA delivered by electrodes attached to the scalp. 1 real sessions of tDCS and 3 sham.
  Other Names: tDCS Minimal Dose
  Arms: tDCS Minimal dose
Device: Sham Transcranial Direct Current Stimulation — Four sessions of sham tDCS; control intervention.
  Other Names: Sham tDCS
  Arms: Sham tDCS

SUMMARY:
The proper control of acute and chronic pain is one of the most important areas in health care. Despite the profound advances in neuroscience over the past 20 years, the investigators still largely use opiate narcotics, much as was done in the Civil War. Total knee arthroplasty (TKA) is one of the most common orthopedic procedures performed 1. While knee pain is often a complaint that precedes TKA, the procedure itself is associated with considerable post-operative pain lasting days to weeks. Adequate postoperative pain control is an important factor in determining recovery time and hospital length of stay. New analgesic strategies are needed that can be used adjunctively to existing strategies with the potential to reduce reliance on opioid analgesia. Several novel brain stimulation technologies including transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS) are beginning to demonstrate promise as treatments for a variety of pain conditions. Electricity has no metabolite or other residue, and can be delivered with minimal discomfort and without problems associated with drug-drug interactions. In two independent preliminary pilot studies, the Investigators have shown that tDCS can reduce post-operative PCA use by as much as 46% while simultaneously reducing subjective pain ratings. The present study aims to determine the effects of transcranial direct current stimulation (tDCS) on post-operative pain, patient-controlled analgesia (PCA) use, and post-surgical complications during the 48-hour post-operative period following total knee arthroplasty.

DETAILED DESCRIPTION:
The proposed study employs a randomized, double-blind, sham-controlled design to evaluate the effects of tDCS on pain among Veterans receiving unilateral total knee arthroplasty (TKA) and unilateral total hip arthroplasty (THA). Further, this study will examine dose-dependency of the tDCS analgesic effects. Each tDCS session delivered either 20 min of real or sham tDCS. Real tDCS was administered at 2mA whereas sham tDCS delivered none.

120 patients undergoing TKA will be randomly assigned to one of four groups:Group 1 will have 4 sessions of real tDCS, Group 2 - 2 sessions of real tDCS (+ 2 sham-sessions), and Group 3 - 1 session of real tDCS (+ 3 sham-sessions). Group 4 is "Sham" tDCS, which does not involve any real stimulation. The participants will receive 2 tDCS treatments on the day of their surgery, and 2 tDCS treatments the day after their surgery.

ELIGIBILITY:
Inclusion Criteria:

Participants will be 120 patients undergoing TKA or THA surgery at the Ralph H. Johnson VAMC in Charleston SC.

* Between the ages of 19 and 90
* Mentally capable of reading, writing, giving consent, and following instructions
* Cleared for and scheduled for unilateral TKA or THA surgery

Exclusion Criteria:

* Implanted medical devices above the waist
* Pregnant
* History of seizures
* Allergic to latex rubber
* Psychiatric conditions other than for depression and/or anxiety disorders

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Borckardt, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS Full Dose: 4 active treatments administered at 2mA for 20minutes each sessions, two the day of surgery and two the day after surgery.
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- tDCS Half Dose: 2 active treatments administered at 2mA for 20minutes each sessions. 2 real sessions the day of surgery and 2 sham sessions the day after surgery.
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- tDCS Minimal Dose: 1 active treatment administered at 2mA for 20minutes for the first session immediately following surgery, then 1 sham session later, day of surgery, and 2 sham sessions the day after surgery.
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- Sham tDCS: no active treatments. All 4 sessions were sham tDCS. 2 delivered day of surgery, 2 delivered day after surgery.
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
Period: Overall Study
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS
Started | 30 | 30 | 30 | 29
Completed | 30 | 30 | 30 | 29
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- tDCS Full Dose: 4 active treatments
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- tDCS Half Dose: 2 active treatments
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- tDCS Minimal Dose: 1 active treatment
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- Sham tDCS: no active treatments
  Transcranial Direct Current Stimulation: Stimulation of brain areas associated with pain perception using low amplitude direct current delivered by electrodes attached to the scalp.
- Total: Total of all reporting groups
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS | Total
Number analyzed (Participants) | 30 | 30 | 30 | 29 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.73) | 67.0 (8.95) | 63.5 (7.93) | 64.2 (8.14) | 64.7 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 7
  Male | 28 | 29 | 27 | 28 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 29 | 29 | 28 | 116
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 10 | 9 | 34
  White | 22 | 22 | 19 | 19 | 82
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 30 | 29 | 119
Procedure Type [Count of Participants; unit: Participants]
  Total Knee Arthroplasty (TKA) | 18 | 21 | 23 | 20 | 82
  Total Hip Arthroplasty (THA) | 12 | 9 | 7 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Pain Medication Dose
Description: Patient Controlled Analgesia pump usage will be measured (mg of morphine-equivalent) during the acute post-operative period.
Time Frame: 2-Days
Measure: Mean (Standard Error); unit: mg of morphine equivalent dose (MED)
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS
Number analyzed (Participants) | 30 | 30 | 30 | 29
mg of morphine equivalent dose (MED) | 26.99 (2.99) | 31.12 (3.73) | 28.65 (31.12) | 33.15 (5.60)

2. Primary Outcome: Patient-reported Pain Intensity Ratings
Description: Patients reported pain intensity using a visual analog scale (VAS) before and after each tDCS session during the 2 day routine postoperative hospital stay. Patients reported pain intensity by marking a line anchored with a minimum of "0- no pain at all" to maximum of "10- worst pain imaginable." Lower values represent a more favorable outcome. This outcome data is the sum of all VAS scores collected before and after each tDCS session during the 2-day hospital stay, thus each participant had a total of 8 VAS scores during the experimental intervention during hospital stay.
Time Frame: 2-Days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS
Number analyzed (Participants) | 29 | 28 | 29 | 27
score on a scale | 5.33 (.44) | 5.59 (.43) | 5.84 (.48) | 5.33 (.56)

3. Secondary Outcome: Patient-reported Average Pain Ratings
Description: Visual analogue scale pain ratings will be collected during the perioperative and post-discharge periods . Visual analogue scale ratings range from 0-10; a blank line is anchored with a 0 and 10 with the following labels: "0- no pain," "10-worst pain imaginable."
Time Frame: 6 Months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS
Number analyzed (Participants) | 16 | 11 | 13 | 9
score on a scale | 3.06 (.46) | 3.45 (.72) | 3.77 (.74) | 4.89 (.59)

ADVERSE EVENTS:
Time Frame: 2-Days during the routine post-operative hospital stay; the duration in which tDCS was delivered.
Arm/Group | tDCS Full Dose | tDCS Half Dose | tDCS Minimal Dose | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02241967/Prot_SAP_000.pdf